## Donor derived cell-free DNA and rejection of kidney allografts

## MINIMAL RISKS AND CONSTRAINTS HUMAN RESEARCH STUDY

Version N°1.1 of 01/03/2020 Protocol code number: ddcfDNA\_study001

Coordinating Investigator: Professor Alexandre Loupy

Department of Kidney Transplantation

Necker Hospital 149 rue de Sèvres 75015 Paris, France Phone: +33 1 53 98 80 00 Fax: +33 1 53 98 79 54

E-mail: alexandre.loupy@aphp.fr

Scientific Director: Doctor Olivier Aubert

Department of Nephrology

Necker Hospital 149 rue de Sèvres 75015 Paris, France Phone: +33 1 44 49 54 38

Fax: +33 1 44 49 42 30 E-mail: olivier.aubert@aphp.fr

Sponsor: OrganX Foundation

Baarerstrasse 6300 Zug, Switzerland

### PROTOCOL SIGNATURE PAGE

## MINIMAL RISKS AND CONSTRAINTS HUMAN RESEARCH STUDY

Protocol code number: ddcfDNA\_study001

Title: "Donor derived cell-free DNA and rejection of kidney allografts "

Version N°1.1 of: 01/03/2020

The research is carried out in accordance with the current version of the protocol, with GCP and with all statutory and regulatory requirements.

| Coordinating Investigator: Pr Alexandre Loupy Department of Kidney Transplantation Necker Hospital Paris, France | Date:///<br>Signature: |
|---|---|
| Scientific Director: Dr Olivier Aubert Department of Kidney Transplantation Necker Hospital Paris, France | Date:///<br>Signature: |
| Sponsor OrganX Foundation Baarerstrasse 6300 Zug,Switzerland | Date:///<br>Signature: |

## 1 SUMMARY

| Full title | Donor derived cell-free DNA and rejection of kidney allografts |
|---|---|
| Coordinating Investigator | Pr Alexandre Loupy |
| Scientific Director (if applicable) | Dr Olivier Aubert |
| Sponsor | Organ X Foundation |
| Scientific justification | Allograft rejection is a major problem worldwide and results in the loss of thousands of transplants every year, with devastating consequences for patients in terms of mortality, morbidity and quality of life. With a prevalence of approximately 20% in the first-year after kidney transplantation, allograft rejection also represents a considerable economic burden for health care systems with the associated downstream cost related to graft failure and return to dialysis. The standard strategy to monitor rejection is based on surveillance of nonspecific functional markers such as serum creatinine level, estimated glomerular filtration rate, proteinuria and circulating donor-specific anti-HLA antibodies (DSA), which lack sensitivity and specificity. The current gold standard for diagnosing allograft rejection is the biopsy which is a potentially harmful, costly and often unnecessary procedure. Recently, one promising non-invasive biomarkers has emerged in various fields such as oncology or gynecology for the monitoring of the patients: the cell-free DNA. In transplantation, donor-derived cell-free DNA (dd-cfDNA) detected in the blood of transplant recipients has been proposed as a noninvasive biomarker for the detection of rejection. However, dd-cfDNA has not been assessed in an unselected and deeply phenotyped population, with the comparison to the conventional parameters including functional, clinical or immunological factors to monitor patients and detect rejection. |
| Main objective and primary endpoint | Main objectives To assess the association of dd-cfDNA with the presence, activity and severity of allograft rejection, and determine whether dd-cfDNA adds value to standard of care monitoring parameters in detecting kidney allograft rejection |

| | Primary endpoint Kidney allograft rejection (all causes) Time Frame: Up to 10 years after kidney transplantation |
|---|---|
| Design of the study | Type of study: Multicenter international study Time Perspective: prospective |
| Population of study participants | <u>Derivation cohort</u> : Prospective cohort of kidney transplant recipients recruited in 2 French centers |
| | <u>Validation cohort</u> : kidney transplant recipients in 11 North-American centers and 1 Belgian center with clinical, biological, histological and immunological data, and dd-cfDNA assessment. |
| Inclusion criteria | <ul> <li>Recipients transplanted from a deceased or living donor, who<br/>undergone a kidney allograft biopsy with clinical, biological,<br/>histological and immunological data. Written informed consent<br/>at the time of transplantation for the center database.</li> </ul> |
| Exclusion criteria | <ul> <li>Combined organ transplantation</li> <li>Pregnant women</li> <li>Bone marrow transplant</li> </ul> |
| Interventions or product under investigation | This study involves minimal risk and constraints. The intervention consists in the evaluation of the risk of allograft rejection based on parameters measured as part of the standard of care and dd-cfDNA. No medicinal product is under investigation in this protocol. |
| Other interventions added by the study | Gene expression measurement in allograft biopsies |
| Expected benefits for the participants and for society | There will be no immediate individual benefit for the patient to participate in the study. This study will be the first that evaluates the independent association of dd-cfDNA with rejection and its added value in addition to conventional features to predict kidney allograft rejection. This first integrative system will improve the patient monitoring and will help physicians in decision-making process. |

| The intervention added by the study represents minimal risk and constraints for the patient as it will be embedded within the standard of care. No additional puncture is performed; only one additional blood tube is taken for the measurement of dd-cfDNA. |
|---|
| Kidney transplantation; non-invasive diagnosis of rejection for improving patient monitoring |
| Number of participants with post-transplant risk evaluation: Derivation prospective cohort: 1000 patients External validation cohort: 1500 patients |
| Multicenter international study involving 14 sites. |
| Derivation cohort: |
| <ul> <li>Saint-Louis Hospital, Paris, France</li> </ul> |
| Necker Hospital, Paris, France |
| Validation cohort: |
| <ul> <li>Leuven Hospital, Leuven, Belgium</li> </ul> |
| Cedars-Sinai, Los Angeles, USA |
| UCLA, Los Angeles, USA |
| Emory University, Atlanta, USA |
| <ul> <li>Intermountain Medical Center Transplant Services, Murray,<br/>USA</li> </ul> |
| Weill-Cornell Medical School, New York, USA |
| New York Hospital Medical Center, New York, USA |
| Virginia Commonwealth University, Richmond, USA |
| Washington University School of Medicine in St. Louis, St. |
| Louis, pediatric department |
| <ul> <li>Washington University School of Medicine in St. Louis, St.<br/>Louis, adult department</li> </ul> |
| <ul> <li>Transplant Institute, Tampa General Hospital, Tampa, USA</li> <li>University of Wisconsin, Madison, USA</li> </ul> |
| Inclusion period 2011- 2022;<br>Participation period (follow-up): Derivation and validation cohorts:<br>up to August 2022 |

# Expected number of enrolments per site

Derivation cohort (n=1000)

External validation cohorts (n=1500)

#### Statistical analysis

Continuous variables will be described using means and standard deviations (SDs) or median and the interquartile range. We will compare means and proportions between groups using Student's t-test, analysis of variance (ANOVA) (Mann-Whitney test for donor specific antibodies (DSA) mean fluorescent intensity) or the chi-square test (or Fisher's exact test if appropriate).

We will evaluate the association between the dd-cfDNA levels and each allograft diagnosis (ABMR, TCMR, Mixed rejection, glomerulitis without rejection, polyomavirus nephritis, fibrosis, borderline changes, no specific lesions). Then, to investigate the association of dd-cfDNA with rejection severity, we will compare the mean dd-cfDNA level according to each active and chronic Banff lesion score (ranked from 0 to 3).

#### Evaluation of the association between dd-cfDNA and rejection

The associations between allograft rejection and clinical, functional, and immunologic factors will be first computed using logistic regression analyses. The factors identified in these analyses will be thereafter included in a final multivariable analysis if the p-value of the Wald test is < 0.1. Multivariable logistic regression analysis will be performed using a stepwise backward elimination until each predictor is associated with allograft rejection with a p-value below 0.05. The internal validity of the final model will be confirmed using a bootstrap procedure, which involves generating 1,000 datasets derived from resampling the original dataset and permitting the estimation of the biased corrected 95% CI and the accelerated bootstrap OR.

#### Assessment of the added value of dd-cfDNA

To evaluate the added value of dd-cfDNA, we will assess the performances of the reference model (including independent standard of care predictors of the final multivariable model) with and without dd-cfDNA to evaluate to risk of rejection. The performances of the models to predict rejection will be evaluated with the use of the accuracy of the model, which will be assessed based on its discrimination ability and calibration performance. For each model, the discrimination ability (i.e., the ability to separate patients with different prognoses) of the final model will be evaluated using Area under the curve (AUC). Calibration (the ability to provide unbiased rejection predictions in groups of similar patients) will be assessed based on a visual examination of the calibration plots.

| | We will follow the TRIPOD (Transparent Reporting of a Multivariable Prediction Model for Individual Prognosis or Diagnosis) statement for reporting multivariable prediction model development and validation. |
|---|---|
| | Sensitivity analyses: We will investigate the independent association of dd-cfDNA with rejection and its added value in predicting rejection in different clinical scenarios (biopsies performed during the first year or after one-year post-transplantation, according to the subtypes of rejection, protocol biopsies or biopsies performed for clinical indication) and according to the patient ethnicity. |
| | We will use R (version 4.1.2, R Foundation for Statistical Computing) and STATA (v17) for the descriptive and prediction analyses. Values of p<0.05 will be considered significant, and all tests will be 2-tailed. |
| Sources of monetary support | The study is funded by the OrganX Foundation |